CLINICAL TRIAL: NCT03971526
Title: Magnetic Resonance Post-contrast Vascular Hyperintensities at 3 T: a New Highly Sensitive Sign of Vascular Occlusion in Acute Ischaemic Stroke
Brief Title: Magnetic Resonance Post-contrast Vascular Hyperintensities at 3 T: a Sensitive Sign of Vascular Occlusion in Acute Ischaemic Stroke
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 29426989
Record Dates: First submitted 2019-05-26; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Acute Ischaemic Stroke
Keywords: Cerebrovascular disorders; Magnetic resonance imaging; Neuroimaging; Prognosis; Stroke
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI images review — MR images were reviewed by one junior radiologist and one senior neuroradiologist, both blinded to clinical, therapeutic and follow-up data.

SUMMARY:
Magnetic resonance imaging (MRI) is the diagnostic cornerstone for precisely identifying acute ischaemic strokes and locating vascular occlusions.

It was observed that a post-contrast three-dimensional turbo-spin-echo T1weighted sequence showed striking post-contrast vascular hyperintensities (PCVH) in ischaemic territories. The aim is to evaluate the prevalence and the meaning of this finding.

This study included 130 consecutive patients admitted for acute ischaemic stroke with a 3-T MRI performed in the first 12 h of symptom onset from September 2014 through September 2016. Two neuroradiologists blinded to clinical data analysed the first MRI assessments.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 and older at onset of an acute ischaemic stroke
* Availability of at least one pre-therapeutic MRI performed in our centre within 12 h of stroke onset, including a post-contrast 3D TSE T1-weighted sequence.

Exclusion criteria:

* Patients with posterior fossa strokes
* Patients with known intracranial vasculitis or MoyaMoya disease
* Presence of severe MR imaging artefacts preventing correct interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 consecutive patients admitted for acute ischaemic stroke with a 3-T MRI performed in the first 12 h of symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
overal survival | 7 years
  from the AR-PML diagnosis date to that of death or censored on 31 December 2015

IPD SHARING:
Plan to Share IPD: No